CLINICAL TRIAL: NCT00626951
Title: The Supreme Laryngeal Mask Airway. A Randomized, Crossover Study With the ProSeal Laryngeal Mask Airway in Paralyzed, Anesthetized Patients
Brief Title: Crossover Study With the ProSeal and Supreme Laryngeal Mask Airway
Acronym: Supreme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Christian Keller MD MSc, Medical University Innsbruck
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 07208763-1
Record Dates: First submitted 2008-02-15; First posted 2008-02-29 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-06

CONDITIONS: Paralysis
Keywords: LMA Supreme; LMA ProSeal; Laryngeal mask airway; Ventilation
MeSH Terms: conditions — Paralysis; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): LMA Supreme
  Interventions: Device: LMA Supreme
- 2 (Experimental): LMA ProSeal
  Interventions: Device: LMA ProSeal

INTERVENTIONS:
Device: LMA Supreme — Extraglottic airway devices
  Arms: 1
Device: LMA ProSeal
  Arms: 2

SUMMARY:
The LMA Supreme is a new extraglottic airway device which brings together features of the LMA ProSeal, Fastrach and Unique. We test the hypothesis that ease of insertion, oropharyngeal leak pressure, fiberoptic position and ease of gastric tube placement differ between the LMA ProSeal and the LMA Supreme in paralyzed anesthetized patients

DETAILED DESCRIPTION:
The LMA Supreme is a new extraglottic airway device which brings together features of both the LMA ProSeal (high seal cuff, gastric access and bite block - to facilitate ventilation, airway protection and airway obstruction, respectively), the LMA Fastrach (fixed cuve tube and guiding handle - to facilitate insertion and fixation) and the LMA Unique (single use - prevention of disease transmission). The new features are that the airway tube incorporates a drain tube within its lumen to shorten and straighten its path, it is oval-shaped to match the shape of the mouth and to reduce rotation in the pharynx, the inner cuff has been strengthened to prevent airway obstruction from infolding and epiglottic fins have been added to prevent airway obstruction from epiglottic downfolding. In the following randomized, crossover study, we test the hypothesis that ease of insertion, oropharyngeal leak pressure, fiberoptic position and ease of gastric tube placement differ between the LMA ProSeal and the LMA Supreme in paralyzed, anesthetized patients

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology physical status grade I-II
* Age 18-80 yr
* Elective gynecological surgery
* Supine position

Exclusion Criteria:

* Known or predicted difficult airway
* Body mass index >35 kg m-2
* Risk of aspiration

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2007-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | 5 min

SECONDARY OUTCOMES:
Ease of insertion | 1 min

CONTACTS AND LOCATIONS:
Overall Officials: Christian Keller, MD, MSc, Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria